CLINICAL TRIAL: NCT07387653
Title: Feasibility and Clinical Utility of Paired Non-Invasive Hemodynamic and Tissue Oximetry Monitoring to Detect Limb Ischemia in Lithotomy-Positioned Surgeries
Acronym: LIMB
Status: Not yet recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Randa Jalloul, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-25-0372
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Neuropathy;Peripheral; Limb Ischemia
Keywords: trendelemberg; nerve injury; position nerve injury; prolonged surgery
MeSH Terms: conditions — Neuritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prolonged Lithotomy Surgery Cohort: Prolonged Lithotomy Surgery Cohort
  Interventions: Other: Lower-Extremity Perfusion Monitoring

INTERVENTIONS:
Other: Lower-Extremity Perfusion Monitoring — This study involves non-interventional physiologic monitoring only, with no alteration to standard surgical or anesthetic care. After induction of anesthesia, patients will have a non-invasive finger cuff applied for continuous beat-to-beat blood pressure and hemodynamic monitoring, along with bilateral lower-leg tissue oximetry sensors placed over the medial calf to continuously measure tissue oxygen saturation (StO₂) throughout surgery. The monitoring data are recorded for observational analysis only, and postoperative limb pain, sensation, and motor function are assessed once in the recovery unit using standardized 5-point Likert scales

SUMMARY:
The LIMB Study is a prospective, observational pilot study evaluating the feasibility of combined non-invasive hemodynamic and lower-limb tissue oximetry monitoring during prolonged minimally invasive pelvic surgeries performed in lithotomy position. Thirty patients will undergo continuous intraoperative monitoring, with the primary outcome being the frequency and duration of tissue oxygen desaturation events and secondary outcomes examining correlations with postoperative limb pain, sensation, and motor function. The study is non-interventional, poses minimal risk, and aims to generate preliminary data to inform future strategies for early detection and prevention of limb ischemia and well-leg compartment syndrome

DETAILED DESCRIPTION:
Well-leg compartment syndrome (WLCS) is a rare but potentially devastating complication associated with prolonged surgical procedures performed in the lithotomy position. Prolonged limb elevation, external compression, and reduced perfusion pressure can lead to muscle ischemia, nerve injury, and long-term functional impairment. Early clinical detection of limb ischemia is challenging in anesthetized patients, as classic signs and symptoms often present late in the disease course. As a result, subclinical ischemic events may go unrecognized until postoperative neurologic or motor deficits are identified.

Near-infrared spectroscopy (NIRS)-based tissue oximetry and continuous non-invasive hemodynamic monitoring have emerged as promising technologies for early detection of tissue hypoperfusion. The Edwards Acumen IQ non-invasive hemodynamic monitoring system provides continuous beat-to-beat blood pressure and derived cardiovascular parameters, while the ForeSight IQ tissue oximetry system provides absolute tissue oxygen saturation (StO₂) measurements without the need for a baseline calibration. These systems are FDA-cleared and currently used in clinical settings such as extracorporeal membrane oxygenation (ECMO), where reductions in tissue oxygenation have been shown to correlate with limb ischemia.

This prospective, observational pilot study is designed to evaluate the feasibility and clinical utility of combining continuous non-invasive hemodynamic monitoring with bilateral lower-extremity tissue oximetry in patients undergoing prolonged minimally invasive pelvic surgery in the lithotomy position. The study is non-interventional, and no changes to intraoperative or postoperative clinical management will be made based on monitoring data.

A total of 30 adult patients undergoing minimally invasive hysterectomy, myomectomy, or endometriosis surgery in lithotomy position with an anticipated operative duration greater than two hours will be enrolled at a single academic medical center. Patients who are pregnant, undergoing open procedures, expected to have surgery lasting less than two hours, or who have a known allergy to medical adhesives will be excluded. No vulnerable populations will be enrolled.

After informed consent is obtained in the preoperative area, patients will undergo standard anesthesia and surgical care. Following induction of anesthesia, bilateral ForeSight IQ tissue oximetry sensors will be placed longitudinally over the medial calf muscles, and an Acumen IQ finger cuff will be applied for continuous non-invasive hemodynamic monitoring. Devices will be calibrated, and baseline hemodynamic and tissue oxygenation values will be recorded prior to surgical positioning. Continuous monitoring will be maintained throughout the intraoperative period.

The primary outcome is the occurrence and duration of intraoperative lower-extremity tissue oxygen desaturation events, defined as either a greater than 15% decrease from baseline StO₂ or an absolute StO₂ value below 50% sustained for more than five minutes. These events will be recorded retrospectively from device output and analyzed descriptively.

Secondary outcomes include the correlation between intraoperative tissue oxygenation changes and postoperative lower-extremity symptoms. In the post-anesthesia care unit (PACU), patients will complete a brief standardized assessment rating limb sensation, pain, and motor function on a 5-point Likert scale prior to discharge. The electronic medical record will be reviewed for up to 30 days postoperatively to identify any documented neurologic or musculoskeletal complications related to lower-extremity perfusion.

Demographic data, surgical characteristics, and known risk factors for limb ischemia will be collected from the electronic health record and stored in a secure REDCap database. Data will be de-identified for analysis, with linkage logs stored separately and securely.

As this is an observational feasibility study, no direct clinical benefit is expected for participants. Risks are minimal and primarily related to potential skin irritation from adhesive sensors. No study-related interventions are performed. Study findings may inform future protocols aimed at early detection and prevention of limb ischemia during prolonged surgeries in lithotomy position.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients
2. Undergoing minimally invasive pelvic surgery (such as hysterectomy, myomectomy, or endometriosis surgery)
3. Surgery performed in lithotomy position
4. Expected surgical duration > 2 hours as determined by the primary surgeon

Exclusion Criteria:

1. Pregnant patients
2. Procedures expected to last < 2 hours
3. Open surgical approaches
4. Minor procedures
5. Known allergy or sensitivity to adhesives used for monitoring sensors
6. Vulnerable populations (incarcerated, elderly or pregnant)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of 30 adult patients undergoing minimally invasive pelvic surgery-including hysterectomy, myomectomy, or endometriosis surgery-performed in the lithotomy position at a single tertiary care center. Eligible patients are those whose procedures are expected to last longer than two hours, placing them at potential risk for lower-limb ischemia related to prolonged positioning. This cohort represents a typical gynecologic surgical population without inclusion of pregnant or other vulnerable individuals
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-29 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
StO₂ desaturation episodes | Duration of the surgery
  Intraoperative lower-limb tissue oxygenation events, defined as the number and duration of StO₂ desaturation episodes, including a drop >15% from baseline or an absolute StO₂ <50% lasting more than 5 minutes, recorded continuously during surgery

SECONDARY OUTCOMES:
Postoperative lower-limb symptoms- Pain | up to 2 hours
  Postoperative lower-limb symptoms assessed in the post-anesthesia care unit using the following rating scale range 1 through 5, the higher the better.
  1. No sensation (completely numb)
  2. Severely reduced sensation
  3. Moderately reduced sensation
  4. Slightly reduced sensation
  5. Normal sensation
Postoperative lower-limb symptoms-Motor | up to 2 hours post surgery
  Rated using the following scale (range 1-5), higher is better,
  1. No movement (complete paralysis)
  2. Severe motor impairment
  3. Moderate motor impairment
  4. Slight motor impairment
  5. Normal movement
Post-operative Limb symptom- sensation | up to 2 hours after surgery
  Using the following scale range 1-5, higher is worst.
  1. No pain
  2. Mild pain
  3. Moderate pain
  4. Severe pain
  5. Worst possible pain

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Hermann Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No